CLINICAL TRIAL: NCT03500198
Title: Clinical Investigation of the Safety and Effectiveness of the Next-Generation TECNIS® Symfony® Intraocular Lens Model ZHR00
Brief Title: Clinical Investigation of the Next Generation Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUR-IOL-652-2001
Record Dates: First submitted 2018-04-09; First posted 2018-04-18 (Actual); Results first posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Investigational Device: Next Generation TECNIS IOL (Experimental): Investigational Intraocular Lens Device #1: Next Generation TECNIS IOL
  Interventions: Device: Investigational Intraocular Lens Device #1: Next Generation TECNIS IOL
- Control Device: TECNIS Monofocal IOL (Active Comparator): Control Monofocal Intraocular Lens: TECNIS Monofocal IOL
  Interventions: Device: Control Monofocal Intraocular Lens: TECNIS Monofocal IOL

INTERVENTIONS:
Device: Investigational Intraocular Lens Device #1: Next Generation TECNIS IOL — Intraocular lens replaces the natural lens removed during cataract surgery.
  Arms: Investigational Device: Next Generation TECNIS IOL
Device: Control Monofocal Intraocular Lens: TECNIS Monofocal IOL — Intraocular lens replaces the natural lens removed during cataract surgery.
  Arms: Control Device: TECNIS Monofocal IOL

SUMMARY:
An investigational IOL designed to provide improved intermediate and near visual acuity and decreased spectacle wear was evaluated for safety and effectiveness in a six-month study.

DETAILED DESCRIPTION:
The next generation TECNIS IOL designed to provide improved intermediate and near visual acuity and decreased spectacle wear was evaluated for safety and effectiveness in a six-month interventional study and compared to a marketed monofocal IOL. Assessments included distance-corrected intermediate and near visual acuity, depth of focus at 0.2 logMAR and spectacle wear frequency.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 22 years of age
* Bilateral cataracts for which posterior chamber IOL implantation has been planned
* Corneal astigmatism:
* Normal corneal topography
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures and study visits
* Signed informed consent and HIPAA authorization or equivalent documentation necessary to comply with applicable privacy laws pertaining to medical treatment in the governing countries
* Ability to understand and respond to a questionnaire in English

Exclusion Criteria:

* Irregular corneal astigmatism
* Inability to focus or fixate for prolonged periods of time (e.g., due to strabismus, nystagmus, etc.)
* Prior corneal refractive (LASIK, LASEK, RK, PRK, etc.) or intraocular surgery, Including prophylactic peripheral iridotomies and peripheral laser retinal repairs
* Poorly-controlled diabetes
* Patient is pregnant, plans to become pregnant, is lactating or has another condition associated with the fluctuation of hormones that could lead to refractive changes
* Concurrent participation or participation within 60 days prior to preoperative visit in any other clinical trial
* Desire for monovision correction

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devi Priya Janakiraman, OD, FAAO, Study Director — Johnson & Johnson Surgical Vision, Inc.
Locations (10):
- United States (10):
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - The Eye Associates of Manatee, LLP, Bradenton, Florida
  - Levenson Eye Associates, Inc., Jacksonville, Florida
  - Jones Eye Clinic, Sioux City, Iowa
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Eye Care Specialists, Kingston, Pennsylvania
  - Vance Thompson Vision Clinic, Prof LLC, Sioux Falls, South Dakota
  - Key-Whitman Eye Center, Dallas, Texas
  - Berkeley Eye Institute, P.A., Houston, Texas
  - Slade & Baker Vision, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 247 participants signed the informed consent form and out of them 27 participants were never randomized and treated, 2 were randomized but not treated. Hence 218 participants were implanted lens in the first eye, (110 in ZHR00 and 108 in ZCB00 control group).
Groups:
- Investigational Device: ZHR00: Investigational next-generation TECNIS foldable intra ocular lens (IOL) designed for placement in the capsular bag were implanted in participants eyes who planned to have bilateral cataract surgery.
- Control Device: ZCB00: TECNIS control monofocal model ZCB00 foldable IOL designed for placement in the capsular bag were implanted in participants eyes who planned to have bilateral cataract surgery.
Period: Overall Study
Arm/Group | Investigational Device: ZHR00 | Control Device: ZCB00
Started | 110 | 108
First Eye | 110 | 108
Second Eye | 109 | 108
Completed | 110 | 107
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat (mITT) population included all eyes randomized and implanted with either a test or control study intraocular lens (IOL) in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Device: ZHR00 | Control Device: ZCB00 | Total
Number analyzed (Participants) | 110 | 108 | 218
Age, Customized [Number; unit: Participants]
  less than < 60 Years | 15 | 13 | 28
  60-69 Years | 49 | 49 | 98
  70-79 Years | 43 | 40 | 83
  Greater than or equal to >= 80 Years | 3 | 6 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 75 | 146
  Male | 39 | 33 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 102 | 105 | 207
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian (including Indian) | 4 | 3 | 7
  Black | 6 | 14 | 20
  Native Hawaiian/Pacific Islander | 0 | 1 | 1
  Caucasian | 99 | 90 | 189
  Other Race | 1 | 0 | 1
  American Indian/Alaska Native | 0 | 0 | 0
  Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Monocular, Photopic Distance Corrected Intermediate Visual Acuity (DCIVA) at 66 Centimeter (cm)
Description: Visual Acuity (VA) was assessed monocularly (each eye separately) under photopic (well-lit) conditions using best distance correction (distance refraction) and high contrast, Early Treatment Diabetic Retinopathy Study (ETDRS) chart at 66 cm from spectacle plane. It was measured in logarithm of the minimum angle of resolution (logMAR), on an ETDRS chart. A lower numeric value represented better VA. This analysis was pre-specified for the first operative eye only.
Time Frame: 6 months (postoperative)
Population: The safety (SF) population included all eyes and subjects implanted in at least one eye with either a test or control IOL with data available at the time of analysis (i.e., no data imputation). Here 'N' (number of participants and number of eyes analyzed) signifies the number of participants and their first eye evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Investigational Device: ZHR00 | Control Device: ZCB00
Number analyzed (Participants) | 110 | 107
Number analyzed (Eyes) | 110 | 107
logMAR | 0.053 (0.149) | 0.370 (0.173)
Statistical Analysis 1: Comparison: Investigational Device: ZHR00 vs Control Device: ZCB00; Test type: Superiority; p < 0.0001, t-test, 1 sided

2. Primary Outcome: Monocular Photopic Distance Corrected Depth of Focus Assessed by the Mean Defocus Curve
Description: Depth of focus was assessed using best corrected distance refraction, and 100% contrast ETDRS letters. VA was measured between +2.00 Diopter (D) and -4.00 D in 0.5 D defocus steps. VA was measured in logMAR. The depth of focus was estimated as the dioptric range between zero defocus and the first point on the negative lens induced mean defocus curve that crosses the 0.2 logMAR using a linear interpolation. A lower numeric value represents better VA. This analysis was pre-specified to be reported for the first operative eye only.
Time Frame: 6 months (postoperative)
Population: as for outcome 1
Measure: Mean (Full Range); unit: diopter
Units Other Than Participants: Eyes
Arm/Group | Investigational Device: ZHR00 | Control Device: ZCB00
Number analyzed (Participants) | 109 | 106
Number analyzed (Eyes) | 109 | 106
diopter | 2.3 [2.1 to 2.6] | 0.8 [0.7 to 1.0]

3. Secondary Outcome: Monocular, Photopic Distance Corrected Near Visual Acuity (DCNVA) at 40 cm
Description: Visual acuity was tested monocularly under photopic conditions using best distance correction (distance refraction) and high contrast, ETDRS chart set at 40 cm from the spectacle plane using the near point rod. VA was measured in logMAR on an ETDRS chart. A lower numeric value represented better VA. This analysis was pre-specified to be reported for the first operative eye only.
Time Frame: 6 months (postoperative)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | Investigational Device: ZHR00 | Control Device: ZCB00
Number analyzed (Participants) | 110 | 106
Number analyzed (Eyes) | 110 | 106
LogMAR | 0.151 (0.148) | 0.466 (0.203)
Statistical Analysis 1: Comparison: Investigational Device: ZHR00 vs Control Device: ZCB00; Test type: Superiority; p < 0.0001, t-test, 1 sided

4. Secondary Outcome: Overall Spectacle Wear
Description: Overall spectacle wear was determined for participants wearing glasses or contact lenses using Patient-Reported Spectacle Independence Questionnaire (PRSIQv2) asking if their response is 'none of the time' in all the 4 conditions (distance vision, intermediate vision, near vision and overall vision) of the spectacle wear questions were reported. PRSIQv2 questionnaire responses were divided into two response groups: reports of "none of the time" and the combined reports of "a little of the time," "some of the time," "most of the time," or "all of the time".
Time Frame: 6 months (postoperative)
Population: The modified intent-to-treat (mITT) population included all eyes randomized and implanted with either a test or control study intraocular lens (IOL) in the study. Here 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Investigational Device: ZHR00 | Control Device: ZCB00
Number analyzed (Participants) | 109 | 108
Percentage of participants | 63.3 | 7.6
Statistical Analysis 1: Comparison: Investigational Device: ZHR00 vs Control Device: ZCB00; Test type: Superiority; p < 0.0001, 1-sided logistic regression

ADVERSE EVENTS:
Time Frame: Up to 11.5 months
Description: The SF population included all eyes and participants implanted in at least one eye with either a test or control IOL with data available at the time of analysis (that is, no data imputation). Adverse events (AEs) were planned to be reported for each eye separately and AEs not related to eyes were counted and represented in both the eyes.
Groups:
- Investigational Device: ZHR00 (First Eye); Investigational Device: ZHR00 (Second Eye): Investigational next-generation tecnis symfony, model ZHR00 foldable intra ocular lens (IOL) designed for placement in the capsular bag were implanted in participants eyes to have cataract surgery using the unfolder platinum 1 series implantation system.
- Control Device: ZCB00 (First Eye); Control Device: ZCB00 (Second Eye): Investigational next-generation tecnis control monofocal model ZCB00 foldable IOL designed for placement in the capsular bag were implanted in participants eyes to have cataract surgery using the unfolder platinum 1 series implantation system.
Arm/Group | Investigational Device: ZHR00 (First Eye) | Control Device: ZCB00 (First Eye) | Investigational Device: ZHR00 (Second Eye) | Control Device: ZCB00 (Second Eye)
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/108 | 0/109 | 0/108
Serious Adverse Events (participants affected / at risk) | 5/110 | 5/108 | 6/109 | 4/108
Other Adverse Events (participants affected / at risk) | 9/110 | 1/108 | 9/109 | 1/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Device: ZHR00 (First Eye) (N=110) | Control Device: ZCB00 (First Eye) (N=108) | Investigational Device: ZHR00 (Second Eye) (N=109) | Control Device: ZCB00 (Second Eye) (N=108)
Retinal Detachment (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Cystoid macular edema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lens dislocation (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypopyon (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cortical Remnant in anterior chamber (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospitalization for vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atherosclerosis with intermittent claudication (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hospitalization for Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Hospitalization for myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Device: ZHR00 (First Eye) (N=110) | Control Device: ZCB00 (First Eye) (N=108) | Investigational Device: ZHR00 (Second Eye) (N=109) | Control Device: ZCB00 (Second Eye) (N=108)
Adverse Device Effects due to visual symptoms (Product Issues) | 9 (9) | 1 (1) | 9 (9) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review results communication prior to public release and can embargo communications regarding trial results at anytime

DOCUMENTS (2):
  • Study Protocol (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT03500198/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT03500198/SAP_001.pdf